CLINICAL TRIAL: NCT06728930
Title: Evaluation of a Novel Microbiological Diagnostic Test for Latent Mycobacterium Tuberculosis Infection
Acronym: MICRO-LTBI
Status: Enrolling by invitation | Type: Observational
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Other Study IDs: 59558
Record Dates: First submitted 2024-10-31; First posted 2024-12-11 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Latent Tuberculosis Infection; Tuberculosis Infection, Latent
Keywords: Tuberculosis; Tuberculosis Infection; Latent Tuberculosis; Latent TB; Diagnosis of latent TB; detection of TB in blood; Mtb detection in blood; TB PCR in blood
MeSH Terms: conditions — Latent Tuberculosis; Tuberculosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Cryopreserved PBMC and heat treated PBMC and lysed cell samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Latent TB screenees: Patients attending TB clinic who are being screened for latent TB. Includes recent migrants from a country with high TB prevalence, occupational health referrals with a positive IGRA, household contacts of TB cases and patients who are about to start biological therapy (eg. anti-TNF)
- Active TB patients: Patients with active TB who are not already on anti-tuberculous treatment

SUMMARY:
Tuberculosis (TB) is an infectious disease that is caused by bacteria (bugs). The infection is passed on when a patient with active lung TB coughs bugs into the air, which are then breathed in by an uninfected person. In 90% of people who get infected, the TB infection remains dormant and the person never falls ill with active TB disease. However, 10% of people with dormant TB infection will eventually go on to develop active TB disease at some time in the future, with symptoms such as cough and weight loss. Dormant TB infection can be treated with a 3-month course of antibiotics, which prevent the infection from becoming active and causing problems in the future. However, existing tests for dormant TB rely on detecting the body's immune response to infection, rather than detecting the TB bugs themselves. Because the immune response doesn't go away when dormant TB is treated, existing tests for dormant TB do not change from positive to negative after antibiotic treatment.

Thus, clinicians can't know if antibiotic treatment of dormant TB infection was successful or not.

Moreover, existing tests can't distinguish the 90% of people with dormant TB infection who will never develop active TB (and who don't need antibiotics) from the 10% who will go on to fall ill with active TB at some point in the future (who do need antibiotics). So the investigators end up giving antibiotics to many more people than we need to. Recently, a group of scientists in Germany have developed a sensitive new blood test that was able to detect very small numbers of TB bugs in the blood of just seven people with dormant TB infection. This finding has created a lot of excitement in the TB field, as nobody has been able to find TB bugs in people with dormant infection before. Our research study will evaluate this new blood test in a larger group of 100 people, with and without dormant TB infection, to see if the findings from Germany are really true. If they are, then this could lead to the development of a more accurate test for dormant TB infection in the future.

DETAILED DESCRIPTION:
Objectives:

i) To determine whether M. tuberculosis (Mtb) DNA can be detected in CD34+ peripheral blood mononuclear cells (PBMC) isolated from

* asymptomatic adults being screened for LTBI (LTBI screenees)
* adults with newly-diagnosed active tuberculosis (active cases) ii) To determine whether strains of Mtb isolated from CD34+ PBMC of recent household TB contacts are genetically identical to those isolated from the sputum of index cases with pulmonary TB to whom they have been exposed iii) To characterise immunological, clinical and epidemiological correlates of ability to detect Mtb in CD34+ PBMC in a heterogeneous population of IGRA-positive and -negative LTBI screenees.

iv) To determine whether presence of Mtb DNA in CD34+ PBMC of IGRA-positive LTBI screenees associates with the presence of a peripheral blood transcriptional signature recently reported to predict risk of progression to active TB v) To assess longitudinal change in CD34+ PCR assay results in

- LTBI screenees completing chemoprophylaxis for LTBI

* LTBI screenees not receiving chemoprophylaxis
* Patients completing treatment for active TB

4.1. Background

Tuberculosis (TB) is an infectious disease caused by organisms of the M. tuberculosis complex (MTBC). The primary pathogen in humans is M.tuberculosis (Mtb). TB commonly affects the lungs and is transmitted through inhalation of infectious droplets expectorated by a patient with active pulmonary TB. Tuberculosis has been a major cause of morbidity and mortality throughout human history. In Europe and North America, a surge in TB cases in the 17th and 18th century was followed by a rapid decline primarily attributed to improved socioeconomic conditions, application of public health measures and isolation of TB patients.1 Towards the end of the 19th century, after the downward trend of TB cases and deaths in Europe and North America, two major events, the discovery of Mtb and X-ray, became key in the diagnosis and management of TB.1 Subsequently, vaccination with M. bovis bacille Calmette-Guérin (BCG) and antibiotic treatment in the first half of the 20th century led to global optimism that TB control and elimination was within reach. However, TB remains a serious public health threat to this day and it is the second leading infectious cause of death globally. 2, 3 According to the 2015 WHO report, an estimated 9.6 million new TB cases (12% of which were HIV co-infected) and 1.5 million deaths (of which 0.4 million were among HIV co-infected people) occurred globally in 2014.4 In addition, one third of the global population is estimated to have latent Mtb infection (LTBI), of whom around 10% will develop active TB in their lifetime.5

Although only 22 low or middle income countries (LMICs) account for 80% of the global burden, TB is still an important disease among immigrant populations in high income countries. In the United Kingdom (UK), reductions in TB incidence achieved in the 20th century have reversed with a 50% increase in TB notifications between 1998 and 2009.6 In 2013, a total of 7,892 TB cases equivalent to an incidence of 12.3 per 100,000 population per year, the highest among high income countries, were reported.7 A high proportion (37.8%) of TB cases in the UK is found in London, where the TB incidence rate is 35.5 per 100,000 population per year; immigrants from India (30%), Pakistan (20%) and Somalia (5%) accounted for the majority of these cases.7

Currently, the key strategies in TB control are accurate and rapid diagnosis of active disease together with effective treatment to interrupt transmission. However, delayed diagnosis is a major challenge facilitating transmission in communities.8 Generally, it takes several months from the onset of symptoms until a TB patient starts treatment. For example, in the UK, nearly a third of pulmonary TB patients start treatment 4 months after onset of symptoms.7 Such long delays, coupled with the large pool of LTBI suggests the need for interventions to identify and treat individuals with LTBI to achieve TB control. Antimicrobial treatment of LTBI (chemoprophylaxis) is effective in reducing risk of reactivation and is routinely implemented in high income, low incidence settings. However, implementation of this policy, particularly in high burden settings, is hampered by the lack of a diagnostic test to identify the sub-set of Mtb-sensitised individuals who are at risk of developing active TB, at whom chemoprophylaxis should be targeted.

Currently, the diagnosis of LTBI is made by detecting an adaptive immune response to Mtb infection, either in vivo (using the tuberculin skin test) or ex vivo (using Interferon-Gamma Release Assays [IGRAs]). This approach, which does not detect Mtb directly, is limited in that it cannot distinguish the 10% of sensitised individuals who are at risk of reactivation (in whom chemoprophylaxis may be of benefit) from the 90% who are immunologically sensitised but who do not progress to active disease (in whom chemoprophylaxis confers no benefit). This latter group is potentially heterogeneous: some may have eliminated the infection, while others may have LTBI but be able to contain it indefinitely.9 Tools to dissect out these possible phenotypes could allow more precise targeting of chemoprophylaxis, but they are currently lacking. In this study, the investigators will investigate whether Mtb can be detected in CD34+ cells isolated from peripheral blood of a) adults being screened for LTBI (LTBI screenees), and b) adults with newly-diagnosed active TB (active cases).

4.2. Rationale for the study

This study builds on a recent observation by one of the co-investigators (Stephen Reece) who was part of a group at the Max Planck Institute for Infection Biology, Berlin, who have detected Mtb DNA in CD34+ long-term repopulating pluripotent hematopoietic stem cells (LTpHSCs) isolated from 100 ml of peripheral blood of seven healthy adults with LTBI (positive IGRA, active TB excluded); Mtb DNA was not detected in LTpHSCs of seven IGRA-negative healthy adults. 10 If this remarkable finding can be replicated in another setting, it could lead to the development of a novel microbiological test ('the CD34+ PCR assay') with several potential applications:

a) to identify individuals who are latently infected with antibiotic-resistant Mtb (allowing selection of an appropriate chemoprophylaxis regimen), b) to monitor efficacy of chemoprophylaxis and interventions designed to prevent acquisition of LTBI, such as vaccines and programmes of micronutrient supplementation, c) to track spreading of particular strains through a population (providing a tool for public health intervention), d) to discriminate between Mtb-sensitised individuals who are at risk of progression to active disease vs. those who are not, allowing chemoprophylaxis to be targeted at populations who may benefit from it, and e) to provide new insights into the immunobiology of LTBI and the pathogenesis of human tuberculosis.

4.3. Hypotheses

i) Mtb DNA can be detected in CD34+ PBMC of asymptomatic IGRA-positive adults and active cases of TB at diagnosis, but not in IGRA-negative adults.

ii) Strains of Mtb isolated from CD34+ PBMC of asymptomatic IGRA-positive TB contacts will be genetically identical to those isolated from the sputum of index cases of pulmonary TB to whom they have been recently exposed.

iii) Ability to detect Mtb DNA in CD34+ PBMC of LTBI screenees associates with IGRA results as well as recognised clinical and epidemiological risk factors for LTBI iv) Ability to detect Mtb DNA in CD34+ PBMC of IGRA-positive LTBI screenees associates with peripheral blood transcriptomic signatures previously defined to be associated with progression to active TB v) Antimicrobial therapy is effective in eliminating Mtb from CD34+ PBMC isolated from individuals with LTBI or active TB in whom it was detectable at baseline; and that results of the CD34+ PCR assay are reproducible on repetition in LTBI screenees who have not received chemoprophylaxis

5. Objectives

5.1. Primary Objective

To determine whether M. tuberculosis (Mtb) DNA can be detected in CD34+ peripheral blood mononuclear cells (PBMC) isolated from

* asymptomatic adults undergoing routine screening for LTBI (LTBI screenees)
* adults with newly-diagnosed active tuberculosis (active cases)

5.2. Secondary Objectives

* To determine whether strains of Mtb isolated from CD34+ PBMC of TB contacts are genetically identical to those isolated from the sputum of index cases with pulmonary TB to whom they have been exposed
* To characterise immunological, clinical and epidemiological correlates of ability to detect Mtb in CD34+ PBMC in a heterogeneous population of IGRA-positive and -negative LTBI screenees.
* To determine whether presence of Mtb DNA in CD34+ PBMC of IGRA-positive screenees associates with the presence of a peripheral blood transcriptional signature recently reported to predict risk of progression to active TB11
* To assess longitudinal change in CD34+ PCR assay results in
* LTBI screenees completing chemoprophylaxis for LTBI
* LTBI screenees not receiving chemoprophylaxis
* patients completing treatment for active TB

Study Design and Study Visits

The investigators will conduct a longitudinal study. Two groups of participants will be recruited: adults being screened for LTBI (LTBI screenees), and patients about to initiate treatment for active TB (active cases). LTBI screenees are those who are being screened for LTBI as part of standard care: they include recent contacts of an infectious index TB case, new entrants from high TB burden countries, health workers undergoing occupational health screening and patients who are about to undergo immunosuppressive therapy. Patients with active TB are those who have been diagnosed with acitve TB who are about to start taking anti-TB therapy.

At baseline (Visit 1), participants who fulfil inclusion criteria and give written informed consent to participate in the study will be asked to provide sociodemographic information including details of age, sex and ethnic origin as well as details of TB exposure history (including specific exposure to participants with active TB enrolled in the study) and other clinically relevant data, all of which will be recorded on a Case Report Form (CRF). An HIV serology test will be performed if this is not already being done as part of routine care. A 120 ml (117 ml if HIV test is already done as part of routine care) blood sample will be collected for IGRA (QFT-Plus), blood culture for Mtb, peripheral blood transcriptome risk signature analysis and the CD34+ PCR assay for Mtb DNA at baseline. IGRA-positive participants in whom active TB has been excluded using clinical evaluation and chest X-ray (part of standard care) will be offered a 3-month course of rifampicin and isoniazid chemoprophylaxis if they fulfil criteria for this therapy (also part of standard care).12

Communication of positive HIV test results will be handled according to the recommendations of the UK National Guidelines for HIV Testing 2008. Positive HIV test results will be communicated in a face-to-face interview with a study doctor, in the presence of a nurse from the Barts Health NHS Trust Genito-Urinary Medicine (GUM) clinic (the local HIV service). Participants who test HIV-positive will be referred to their nearest GUM clinic for confirmation of their results and further management as appropriate.

At 3 months (Visit 2), details of prescription of and adherence to chemoprophylaxis will be recorded, and a second blood sample (117 ml) will be taken for repeat IGRA (QFT-Plus), blood culture and CD34+ PCR assay. For participants who took chemoprophylaxis, a Tempus tube will also be taken at Visit 2.

At baseline (Visit 1), participants who fulfil inclusion criteria and give written informed consent to participate in the study will be asked to provide basic sociodemographic information including details of age, sex and ethnic origin as well as duration of their symptoms, contact with any enrolled LTBI screenee and other clinically relevant data, all of which will be recorded on a CRF. HIV serology, full blood count and, sputum smear microscopy and cutlure for M.tuberculosis are performed as part of routine care in this patient group. A 114 ml blood sample will be collected for IGRA (QFT-Plus), blood culture for Mtb and the CD34+ PCR assay for Mtb DNA at baseline. TB patients will be treated for active disease according to UK guidelines. 12

Following completion of chemotherapy (Visit 2, usually at 6 months), details of prescription of and adherence to anti-TB treatment will be recorded and a second blood sample (114 ml) will be collected for IGRA (QFT-Plus), blood culture for Mtb and the CD34+ PCR assay.

Study Procedures

Invitation and informed consent procedures

Invitation

In London, screening for LTBI using an IGRA is commonly performed in four groups: recent contacts of active TB patients; new entrants from high TB burden countries; patients who are about to start immunosuppressive therapies; and health workers undergoing occupational health screening. Groups at risk of LTBI may initially be identified in various different settings (TB clinic, primary care, rheumatology clinics, occupational health services), but they are all referred either to a TB clinic (contacts, new entrants, patients about to start immunosuppressive therapy) or to the Occupational Health Clinic (health workers undergoing occupational health screening) for LTBI screening to be performed. Potentially eligible LTBI screenees will therefore be identified and recruited to the study at TB clinics or the Occupational Health Clinic. Patients with active TB will be identified and recruited at Barts Health NHS Trust TB Clinics.

Potentially eligible individuals will be informed about the study by nurses or doctors working in TB clinics or Occupational Health clinic, who perform TB screening as part of usual clinical care.. Those who express an interest in the study will be provided with a Participant Information Sheet by a member of the clinical care team. This will explain the aims, methods, anticipated benefits and potential hazards of the study, and will be presented in non-technical language either in English or other languages where necessary. Those taking a Participant Information Sheet will be asked to complete a 'Contact Slip' providing their contact details and authorising the research team to make contact with them once they have had a chance to read the information; this 'Contact Slip' will be forwarded to the research team by the participant's usual care team.

Informed Consent Procedures

Informed consent will be conducted according to JRMO standard operating procedures. Informed consent will be taken in a private room by personnel who have received specific training in Good Clinical Practice and taking of informed consent, who may be doctors, nurses or research assistants. During the consent process, participants will be advised that participation is voluntary and that they can refuse to enter the study or withdraw at any time during follow-up, for any reason.

Participants will be asked to indicate their consent to participate by signing and printing their name. An impartial witness will be required to countersign consent for those who require an interpreter during the consent process. Participants will be financially compensated for travel expenses associated with each visit.

Enrollment and follow-up procedures

Recruitment at baseline

Potential participants will be assessed for eligibility based on the inclusion and exclusion criteria stated above. Following the consent process and after a participant gives written informed consent to participate, a unique ID number will be assigned. Assessment of eligibility to participate will be performed by suitably trained personnel who may be doctors, nurses or research assistants.

Data collection procedure

Using a CRF, at Visit 1 (V1), all participants will be asked to give sociodemographic information and medical history including medication history. LTBI screenees will be asked to provide details of recent and previous exposure to TB patients, history of TB and other potential determinants of LTBI such as physical proximity to active TB patients, average daily duration of exposure as well as total duration of exposure to index cases. CRFs will also include the following data: checklist of eligibility criteria, results of baseline clinical examinations and laboratory tests, and information collected during follow-up including withdrawal details, if applicable. The members of the project team responsible for completing CRFs, who may be research fellows or field workers, will be listed in a delegation log.

Baseline sample collection and laboratory assessments

Samples will be collected as detailed in Figure 1 and Tables 1 and 2, and laboratory analyses will be perfomed as detailed in Tables 3 and 4. Where tests are performed as part of routine care (e.g. full blood count for patients with active TB, HIV serology for patients with active TB and IGRA-positive LTBI screenees), results will be accessed via CRS and documented on the CRF. IGRA-negative LTBI screenees and unexposed participants will be offered a HIV test at Visit 1.

To investigate whether Mtb strains isolated from CD34+ PBMC of TB contacts match those isolated from sputum of index cases to whom they have been exposed, sputum samples will be collected from 10 index active TB patients who have CD34+ PCR assay positive contacts enrolled in the study, and whole genome sequencing analysis will be performed on isolates cultured from these samples. Based on this analysis, primers to create Mtb amplicon libraries will be designed using bioinformatic approaches to capture strain diversity. These primers will then be used to generate Mtb amplicon libraries from CD34+ cells harbouring Mtb genomic DNA isolated from TB contacts. These libraries will then be sequenced and compared to the Mtb genome of the index case to determine whether strains isolated from index cases and contacts match.

Participants with positive HIV tests / IGRAs will be referred to HIV / TB clinics respectively for further assessment. Where HIV tests and IGRAs have been performed for research purposes (i.e. where they are not part of routine care), research staff will communicate these results to participants when they become available.

Follow-up procedures

* LTBI screenees: Visits and follow-up assessments are detailed in Figure 1, Table 1 and Table 3. Participants will attend visit 2 at 3 months (visit 2, V2). Participants who have completed chemoprophylaxis will have a routine clinical evaluation upon completion of their treatment. Those who do not take chemoprophylaxis will also be followed up at 3 months after V1. In addition to completing a CRF detailing symptoms of active TB (all participants) and adherence to chemoprophylaxis (those receiving chemoprophylaxis), a 117 ml blood sample will be collected for immunological and molecular analysis as detailed in section 13.3 below. On completion of the second visit, participation in the study will end.
* Patients with active TB: Visits and follow-up are detailed in Figure 1, Table 2 and Table 4. Participants taking anti-TB treatment will have a routine clinical evaluation upon completion of their treatment and a second 114 ml blood sample will be collected during this visit for immunological and molecular analysis as detailed in section 13.3 below. Upon completing the second visit, participation in the study will end.

Results of the CD34+ PCR test will not be used to guide clinical management, as this test is a research tool in the early phases of development, and its results have not been correlated with any clinical outcome.

Participant withdrawal

Participants will be withdrawn if they withdraw their consent to participate or if it is concluded that withdrawal is in the participant's best interests. Participants will also be considered to have withdrawn if they fail to attend their second scheduled study visit despite written and telephone reminders. If a participant withdraws from the study, the reason for withdrawal will be recorded in the CRF.

Data collected up to the time of withdrawal will be included in study analyses, unless otherwise requested by a participant. Any clinical samples taken prior to a participant's withdrawal will be used for study analyses.

End of Study Definition

The study will end when all clinical and laboratory assessments are complete for all participants attending follow-up.

9. Statistical Considerations

9.1 Sample size

The main aim of this study is to validate and extend findings from another setting in which genomic DNA of Mtb was detected in CD34+ cells isolated from the peripheral blood of seven IGRA-positive asymptomatic adults.10 To address this objective, a total of 100 LTBI screenees will be recruited to the cross-sectional study (20 participants per independent variable to be tested in the regression analysis). It is anticipate that approximately fifty of these participants will be IGRA-positive, of whom approximately forty will be prescribed chemoprophylaxis: follow-up of 25 of these participants will give >80% power at the 5% significance level to demonstrate a reduction in the proportion of CD34+ PCR-positive individuals from 80% at baseline to 30% at follow-up.

10. Ethical Considerations

Before the start of the study, approval will be sought from the NHS REC for the study protocol, informed consent forms and other relevant documents. The study will not commence until necessary approvals are obtained from the ethics committee and a 'green light' is given to activate sites by the sponsor. The CI will ensure that this study is conducted in accordance with the Declaration of Helsinki (2013) and the ethical principles in the Research Governance Framework for Health and Social Care, Second Edition, 2005 and its subsequent amendments. Decisions as to whether an amendment constitutes a minor or substantial amendment will lie with the sponsor. Substantial amendments that require review by the REC will not be implemented until they are approved by the relevant body. All correspondence with the Sponsor and the REC will be retained in the study Master File. The CI will notify the REC and the Sponsor at the end of the study.

Written informed consent will be obtained from participants by a suitably trained person (who may be a doctor, a nurse or a research assistant) prior to participation in this study. Information sheets will be made available in English and other languages where necessary. Potential participants will be provided with the information sheet and the aims, methods, anticipated benefits and potential hazards of the study will be explained. During the consent process, participants will be explained that participation is voluntary and they can refuse to enter the study or withdraw at any time during follow-up, for any reason.

Conflict of interest

No financial or other competing interests have been identified for the CI or any co-investigator.

11. Safety Considerations

Since the study is observational, the risk of study-related adverse events is negligible. However, any adverse event that is deemed to be related to the study will be reported to the sponsor within 24 hours. The blood volume to be collected (up to 120 ml) may be perceived as large by some participants but adults donating blood commonly give 500 ml at a time without suffering anaemia. The investigators do not therefore anticipate any adverse event related to drawing this volume of blood. Information regarding the volume of blood sample and whether this will have any unwanted health consequences will be explained to participants in the information sheet. All TB patients will be screened for anaemia as part of their usual clinical care and those with haemoglobin level below 10 g/dl at entry will be excluded. In addition, the following measures will be taken to minimise potential inconvenience, discomfort and risk that participants may experience during the course of this study:

- use of suitably trained staff to perform phlebotomy

12. Data Handling and Record Keeping

12.1. Confidentiality

Protected Health Information (PHI) necessary for the conduct and analysis of the study will be collected for all participants screened for the study; this information will include each participant's name, date of birth, sex, address, telephone number, medical record number if applicable, email address if applicable, and ethnic origin. Study staff requiring access to PHI in order to conduct or analyse the study will be listed on a delegation log. PHI will remain confidential, and will be handled, processed, stored and destroyed according to the Data Protection Act 1998. Participants will retain the right to revoke their authorisation for the use of their PHI at any time during the study. All participants will be anonymised in publications arising from this study. Data will be pseudo-anonymised as follows. PHI will be held in a secure database linked to a unique identification code. Clinical information will be held in a separate secure database, linked to the same unique identification code. The CI and co-investigators will have access to the pseudo-anonymised final study dataset.

During the course of research, all records will be the responsibility of the CI and will be kept in secure conditions. When the study is complete, it is the sponsor's requirement that records and data are kept for a further 20 years. The CI will act as the 'Custodian' of the research data. Access to PHI will be limited to the minimum number of individuals necessary for conduct of the study, quality control, audit, and analysis. The following will comprise source documents: screening logs, informed consent and paper CRF. All source documents will be stored securely in locked filing cabinets. Data transfer and transport will be conducted in accordance with the UK Data Protection Act 1998. Person-identifiable information will not be stored, transported or sent to or from any portable device unless that device is encrypted.

12.2. Data Collection, Recording and Handling

Signed consent forms and paper documents containing source data will be securely stored. Study data will be entered onto a database in EpiData Entry software. Staff will receive appropriate training to use the database for data entry. Laboratory data will be entered into the database.

The CI and co-investigators will have access to study data during the study. Study staff who require such access in order to conduct the study will also be given such access as is necessary. Access to study data during the study will also be granted to authorised representatives from the Sponsor, host institution and the regulatory authorities as is necessary.

12.3. Quality Control and Quality Assurance

Study documentation will be made available to representatives of the Sponsor and the REC for quality control and quality assurance as requested.

13. Laboratories

13.1. Sample collection, labelling and processing

Blood samples will be collected by study staff, labelled with participant ID and dated. Tempus tubes will be vigorously shaken immediately after collection according to the manufacturer's recommendations. Samples for blood culture and HIV serology will be transported to Central Laboratories for processing. Remaining blood samples will be transported to The Blizard Institute, where the sample receipt date and time as well as the sample condition (eg. non-clotted) will be recorded in a laboratory log. Samples for the QFT-Plus test will be incubated at 37 °C shortly after receipt of samples for 18 hours, prior to centrifugation and aspiration of supernatants which will be stored at -80C pending analysis for IFN-gamma concentration. Blood samples in Tempus tubes will be stored at -80 °C in a labelled rack pending transport to the Division of Infection and Immunity, University College London for RNA extraction and gene expression profiling. PBMC will be separated from the remaining sample (100 ml), with subsequent isolation of CD34+ cells using magnetic bead sorting. Purity of CD34+ cells isolated will be checked by flow cytometry.

ELIGIBILITY:
i) For LTBI screenees

Inclusion Criteria:

* Age ≥16 years
* Undergoing screening for LTBI
* Gives written informed consent to participate

Exclusion Criteria:

* Known HIV infection
* Declines HIV testing
* Previous antimicrobial treatment for active TB or latent TB infection
* Clinical suspicion of active TB
* Already initiated chemoprophylaxis

ii) For adults with active TB Inclusion criteria

* Age ≥16 years
* Newly-diagnosed active TB about to initiate treatment
* Gives written informed consent to participate

Exclusion criteria

* Known HIV infection
* Declines HIV testing
* Already initiated anti-TB treatment
* Haemoglobin concentration <10 g/dl at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Two groups of participants will be recruited: adults being screened for LTBI (LTBI screenees), and patients about to initiate treatment for active TB (active cases). LTBI screenees are those who are being screened for LTBI as part of standard care: they include recent contacts of an infectious index TB case, new entrants from high TB burden countries, health workers undergoing occupational health screening and patients who are about to undergo immunosuppressive therapy. Patients with active TB are those who have been diagnosed with active TB who are about to start taking anti-TB therapy.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Mtb DNA in blood | 3 years
  Prevalence of Mtb DNA in blood of latent screenees and active TB participants

CONTACTS AND LOCATIONS:
Locations (1):
- Blizard Institute, Queen Mary University London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided